CLINICAL TRIAL: NCT03707509
Title: A Phase III, Randomized, Double-Blind, Multi-center Study to Investigate the Efficacy and Safety of Camrelizumab+Gemcitabine+Cisplatin Versus Placebo+Gemcitabine+Cisplatin in Subjects With Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: Phase III Study of Camrelizumab in Combination With Chemotherapy in Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1210-III-308
Record Dates: First submitted 2018-09-25; First posted 2018-10-16 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; PD-1 Antibody; Cisplatin; Gemcitabine
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; Gemcitabine; Injections; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab + Gemcitabine + Cisplatin (Experimental): subject will receive camrelizumab 200mg every 3 weeks, cisplatin 80mg/m2 on Day 1 of each 21 day, at most 6 cycles, gemcitabine 1000mg/m2, Day 1 and Day 8 of each 21 day, maximum 6 cycles
  Interventions: Drug: Camrelizumab; Drug: Gemcitabine; Drug: Cisplatin
- Placebos + Gemcitabine + Cisplatin (Active Comparator): subject will receive placebos every 3 weeks, cisplatin 80mg/m2 on Day 1 of each 21 day, at most 6 cycles, gemcitabine 1000mg/m2, Day 1 and Day 8 of each 21 day, maximum 6 cycles
  Interventions: Drug: Placebos; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Camrelizumab — Maximum 6 cycles for combined therapy. Camrelizumab maintenance.
  Other Names: SHR-1210
  Arms: Camrelizumab + Gemcitabine + Cisplatin
Drug: Placebos — Maximum 6 cycles for combined therapy.
  Other Names: Placebo - Concentrate
  Arms: Placebos + Gemcitabine + Cisplatin
Drug: Gemcitabine — Maximum 6 cycles for combined therapy.
  Other Names: Gemcitabine Hydrochloride for Injection
Drug: Cisplatin — Maximum 6 cycles for combined therapy.
  Other Names: Cisplantin Injection

SUMMARY:
This study is a randomized, placebo-controlled, double-blind, multicenter phase III clinical study. Target population is patients with recurrent/metastatic nasopharyngeal carcinoma who had not received systemic chemotherapy. Study objective is to compare the efficacy and safety of camrelizumab in combination with gemcitabine and cisplatin with placebo in combination with gemcitabine and cisplatin in study population in China. camrelizumab is a humanized anti-PD1 IgG4 monoclonal antibody.

DETAILED DESCRIPTION:
In this study, eligible subject will be randomized into study arm or control arm to accept study treatment. Treatment cycles of chemotherapy will be at most 6 weeks which will be decided by investigators. Progression-free survival (PFS) determined by the Independent Review Committee (IRC) will be the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤75 years;
2. Subjects with histopathological diagnosis of nasopharyngeal carcinoma;
3. Primarily metastatic (stage IVB as defined by the International Union against Cancer and American Joint Committee on Cancer staging system for NPC, eighth edition) or recurrent NPC that is not amenable for local regional treatment or curative treatment;
4. Has not received prior systemic treatment;
5. Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status
6. Subject must have a measurable target lesion based on RECIST v1.1;

Exclusion Criteria:

1. Allergic to monoclonal antibodies, any camrelizumab components, gemcitabine, cisplatin and other platinum drugs;
2. Prior therapy as follow:

   * Anti-PD-1 or anti-PD-L1;
   * Received last dose of anticancer therapy (including chemotherapy, radiotherapy, targeted therapy, etc.) within 4 weeks of the first dose of study medication;
   * Concurrent medical condition requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment. Except: inhalation or topical corticosteroids. Doses > 10 mg/day prednisone or equivalent for replacement therapy;
   * Received major operations or serious injuries within 4 weeks of the first dose of study medication;
3. Not recovered to ≤CTCAE 1 from adverse events (except for hair loss) due to a previously anti-tumor treatment;
4. Pregnancy or breast feeding;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 24 month
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the Independent Review Committee according to RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free survival | up to 24 month
  Progression-free survival (PFS) assessed by investigators according to RECIST V 1.1
Objective Response Rate (ORR) | up to 24 month
  The percentage of patients with CR and PR assessed by investigators according to Recist v 1.1
Disease Control Rate (DCR) Disease Control Rate (DCR) | up to 24 month
  The proportion of patients who have achieved complete response， partial response and Stable disease assessed by investigators according to Recist v 1.1
Duration of Response (DoR) | up to 24 month
  According to Recist v 1.1 accessed by investigators
2 years Overall Survival (OS) rate | up to 24 month
  The percentage of patients overall survival in 2 years
Adverse Events (AEs) | up to 24 month
  All adverse event/Serious adverse event that occurred during the study period according to CTCAE v 4.03

OTHER OUTCOMES:
Antidrug Antibodies (ADAs) | up to 24 month
  To evaluate the incidence and titers of ADAs against camrelizumab

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Cancer Center of Sun-Yat Sen University (CCSYSU); Qing Yang, MD, Study Director — Jiangsu HengRui Medicine Co., Ltd.
Locations (1):
- Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Y, Sun D, Zhou H, Zhou T, Qu S, Li J, Hu C, Xu M, Li W, Shen L, Wu H, Lang J, Hu G, Luo Z, Fu Z, Qu S, Feng W, Chen X, Lin S, Xie B, Li X, Sun Y, Lin Z, Lin Q, Lei F, Long J, Hong J, Huang X, Zeng L, Wang P, He X, Zhao S, Chen G, Zhang Y, Zhao Y, Fang W, Huang C, Li X, Hong S, Zhang L, Yang Y. Five-Year Outcome of Camrelizumab Plus Chemotherapy in Recurrent or Metastatic Nasopharyngeal Carcinoma: A Secondary Analysis of the CAPTAIN-1st Randomized Clinical Trial. JAMA Oncol. 2026 Jan 29:e256245. doi: 10.1001/jamaoncol.2025.6245. Online ahead of print. PMID 41609753
- [Derived] Xiao BJ, Sima XX, Chen G, Gulizeba H, Zhou T, Huang Y. Predictive and prognostic role of early apolipoprotein A-I alteration in recurrent or metastatic nasopharyngeal carcinoma patients treated with anti-PD-1 therapy. Cancer Med. 2023 Aug;12(16):16918-16928. doi: 10.1002/cam4.6321. Epub 2023 Jul 6. PMID 37409613
- [Derived] Yang Y, Qu S, Li J, Hu C, Xu M, Li W, Zhou T, Shen L, Wu H, Lang J, Hu G, Luo Z, Fu Z, Qu S, Feng W, Chen X, Lin S, Zhang W, Li X, Sun Y, Lin Z, Lin Q, Lei F, Long J, Hong J, Huang X, Zeng L, Wang P, He X, Zhang B, Yang Q, Zhang X, Zou J, Fang W, Zhang L. Camrelizumab versus placebo in combination with gemcitabine and cisplatin as first-line treatment for recurrent or metastatic nasopharyngeal carcinoma (CAPTAIN-1st): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2021 Aug;22(8):1162-1174. doi: 10.1016/S1470-2045(21)00302-8. Epub 2021 Jun 23. PMID 34174189